CLINICAL TRIAL: NCT04849897
Title: Virtual Reality Guided Imagery for Chronic Pain
Acronym: VRGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Limbix Health, Inc. (Industry); BehaVR LLC (Industry)
Responsible Party: Principal Investigator, Steven Richeimer, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS 1900549
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Complex Regional Pain Syndromes; Back Pain
MeSH Terms: conditions — Complex Regional Pain Syndromes; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Comparator: Audio Only Guided Imagery Audio Recordings of Guided Imagery via tablet (Active Comparator): Listen to narrative scripts based on traditional GI audio recordings. The narrative scripts will include psychoeducation content that explains how the mind and brain can influence physical pain and how they can be trained to effect changes in experienced chronic pain. Narration will guide users in breathing and relaxation exercises and explain how patients can continue to exert control over their pain outside of the GI experience.
  Interventions: Other: Active Comparator: Audio Only Guided Imagery
- Experimental: Virtual Reality Guided Imagery Platform and VR Headset (Experimental): VR headset for guided imagery with audiovisual computer-generated VR content to accompany the GI narration. The narrative scripts will include psychoeducation content that explains how the mind and brain can influence physical pain and how they can be trained to effect changes in experienced chronic pain. Narration will guide users in breathing and relaxation exercises and explain how patients can continue to exert control over their pain outside of the VR-GI experience.
  Interventions: Device: Experimental: Virtual Reality Guided Imagery

INTERVENTIONS:
Device: Experimental: Virtual Reality Guided Imagery — Platform and VR Goggles
  Arms: Experimental: Virtual Reality Guided Imagery Platform and VR Headset
Other: Active Comparator: Audio Only Guided Imagery — Audio Recordings of Guided Imagery via an iPAD
  Arms: Active Comparator: Audio Only Guided Imagery Audio Recordings of Guided Imagery via tablet

SUMMARY:
To assess treatment with an at-home Virtual Reality Guided Imagery (VR-GI) intervention, 36 patients with chronic pain (18 with chronic back pain, CBP, and 18 with complex regional pain syndrome, CRPS) will complete a 2-week intervention with at-home daily practice of VR-GI (n = 24) or audio-only GI (n = 12). Pre-post treatment measures of pain intensity, opioid use, functional outcomes, and mood will be collected. Intervention feasibility and patient satisfaction will be evaluated post-treatment via questionnaire and qualitative interview.

DETAILED DESCRIPTION:
○ Chronic pain affects over 100 million adults in the US, resulting in disability, loss of work productivity, and overall reductions in health, making chronic pain a major public health problem with an economic burden estimated at $560-635 billion annually. Opioids, the most frequently prescribed class of drugs to control pain, lack evidence supporting their long-term efficacy and carry a 15-26% risk of misuse and abuse among pain patients, highlighting a critical need to develop effective non-pharmacological interventions for pain. Guided imagery (GI), a cognitive-behavioral technique for guiding patients to create multisensory, imagined scenes to increase well-being, is an effective non-pharmacological intervention for reducing pain. However, its effectiveness is limited by patients' imaging abilities. The long-term objective of this project is to reduce chronic pain and opioid use by developing an at-home virtual reality (VR)-GI intervention to improve chronic pain management using the Limbix VR Kit. Given the enhanced immersiveness and interactivity of VR, VR-GI is expected to reduce pain and reliance on opioids, as well as improve functional outcomes and mood, compared to traditional audio-only GI and usual care. The specific aims are to evaluate feasibility and usability of an at-home VRGI intervention in a 2-week clinical trial. Two 15-min VR-GI experiences that guide patients through psychoeducation, relaxation exercises, and interactive virtual worlds that allow them to control their experience of pain will be evaluated. To assess feasibility of an at-home VR-GI intervention, 36 patients with chronic pain (18 with chronic back pain, CBP, and 18 with complex regional pain syndrome, CRPS) will complete a 2-week intervention with at-home daily practice of VR-GI (n = 24) or audio-only GI (n = 12). Pre-post treatment measures of pain intensity, opioid use, functional outcomes, and mood will be collected. Intervention feasibility and patient satisfaction will be evaluated post-treatment via questionnaire and qualitative interview. This research directly addresses the need to improve pain treatment to prevent opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient at the University of Southern California Pain Center
* - English Fluency
* Diagnosis of chronic back pain or complex regional pain syndrome
* Average pain intensity of 5 on a 0 to 10 scale for more than 3 month
* Access to a device with video and audio capability and sufficient WiFI to participate in on-line sessions

Exclusion Criteria:

* History of significant motion sickness
* Active nausea/vomiting
* Epilepsy
* Significant movement problems
* Significant vision or hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Richeimer, MD, Principal Investigator — Keck School of Medicine, Dept. of Anesthesiology
Locations (1):
- USC Pain Center, Keck School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 96 applicants were recruited, 81 met inclusion criteria. 36 participants were enrolled.
Groups:
- Virtual Reality Guided Imagery (VR-GI): VR headset for guided imagery with audiovisual computer-generated VR content to accompany the GI narration. The narrative scripts will include psychoeducation content that explains how the mind and brain can influence physical pain and how they can be trained to effect changes in experienced chronic pain. Narration will guide users in breathing and relaxation exercises and explain how patients can continue to exert control over their pain outside of the VR-GI experience.
- Audio Only Guided Imagery (AO-GI): Listen to narrative scripts based on traditional GI audio recordings. The narrative scripts will include psychoeducation content that explains how the mind and brain can influence physical pain and how they can be trained to effect changes in experienced chronic pain. Narration will guide users in breathing and relaxation exercises and explain how patients can continue to exert control over their pain outside of the GI experience.
Period: Overall Study
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Started | 24 | 12
Completed | 21 | 11
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Audio Only Guided Imagery (AO-GI) | Virtual Reality Guided Imagery (VR-GI) | Total
Number analyzed (Participants) | 12 | 24 | 36
Age, Customized [Count of Participants; unit: Participants]
  age greater than 18 | 12 | 24 | 36
Sex: Female, Male [Count of Participants; unit: Participants] — binary
  Participants
    Female | 10 | 16 | 26
    Male | 2 | 8 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 11 | 19 | 30
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 18 | 27
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Recruited But Not Enrolled as Documented in Participant Log
Description: Participant log tracks number of recruited participants who are ineligible to participate and/or decline to enroll
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Total Recruited: Recruited participants who are ineligible to participate and/or decline to enroll
Arm/Group | Total Recruited
Number analyzed (Participants) | 96
Participants | 60

2. Primary Outcome: Number of Enrolled Participants Who do Not Complete the Study as Documented in Log
Description: Participant log tracks the number of enrolled participants who discontinue intervention, are lost to follow-up and/or experience adverse events.
Time Frame: Baseline to 2 week follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Number analyzed (Participants) | 24 | 12
Participants | 3 | 1

3. Primary Outcome: Number of Practice Sessions Completed by Participants as Documented in Spread Sheet
Description: Spread sheet documenting proportion of at-home daily GI practice completed over 2-week intervention
Time Frame: Baseline to 2 week follow up
Population: For the VR-Gi group, 23 participants were analyzed as one participant did not receive allocated intervention.
Measure: Mean (Standard Deviation); unit: Daily ratings completed
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Number analyzed (Participants) | 23 | 12
Daily ratings completed | 10.8 (3.58) | 11.4 (4.27)

4. Primary Outcome: Pain Assessed by Pain Numeric Rating Scale
Description: Numeric Rating Scale of self-reported highest, lowest, and average pain scores (0-10) over the last 7 days. Higher scores indicate worse pain outcomes.
Time Frame: Baseline to 2 week follow up
Population: For the VR-GI group, 23 participants were analyzed as one participant did not receive allocated intervention. For the AO-GI group, 11 participants were analyzed as one participant did not complete post-intervention questionnaires.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Number analyzed (Participants) | 23 | 11
units on a scale
  Change in Lowest Score Follow up Baseline | 0.381 (1.36) | 0.091 (1.04)
  Lowest Score Baseline | 4 (1.82) | 3.92 (1.51)
  Lowest Score Follow up | 3.71 (1.95) | 3.64 (1.63)
  Change in Highest Score Follow-up-Baseline | 0.619 (.973) | 0.100 (1.37)
  Highest Score Baseline | 8.42 (0.83) | 7.75 (1.36)
  Highest Score Follow-up | 7.86 (1.01) | 7.4 (0.97)
  Change in Average Score Follow-up-baseline | 0.524 (1.08) | 0.182 (1.08)
  Average Score Baseline | 6.08 (1.18) | 5.75 (1.42)
  Average Score Follow-up | 5.62 (1.5) | 5.46 (1.44)

5. Primary Outcome: Opioid Medication Usage Assessed by Frequency of Use Log
Description: Log with list of medications taken, dosages and frequency of use. Lower frequency indicates better outcomes.
Time Frame: Baseline to 2 week follow up
Population: For the VR-GI group, 3 participants were analyzed as others did not have opioid usage. For the AO-GI group, 4 participants were analyzed as others did not have opioid usage.
Measure: Number; unit: Count of Participants with Reduced Opioi
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Number analyzed (Participants) | 3 | 4
Count of Participants with Reduced Opioi | 0 | 1

6. Primary Outcome: Non-opioid Pain Medication Usage Assessed by Frequency of Use Log
Description: Log with list of non-opioid pain mediction taken, dosages and frequency of use. Lower frequency of use indicates better outcomes
Time Frame: Baseline to 2 week follow up
Measure: Number; unit: Pt. count reduced non-opoid pain med use
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Number analyzed (Participants) | 23 | 11
Pt. count reduced non-opoid pain med use | 6 | 3

7. Secondary Outcome: Anxiety Assessed by Generalized Anxiety Disorder Assessment: GAD-2 (GAD-7)
Description: Generalized Anxiety Disorder Assessment is calculated by assigning scores of 1,2,3 and 4, to the response categories of Not at all sure, Several Days,Over half the days, Nearly every day , respectively. Total score for the two ranges from 0-6 with higher number indicating worse anxiety outcome.
Time Frame: Baseline to 2 week follow up
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on GAD-2 scale
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Number analyzed (Participants) | 23 | 11
score on GAD-2 scale
  Change in GAD (Follow up-Baseline | -1.2 (1.20) | -.06 (1.17)
  GAD Baseline | 1.83 (1.86) | 1.58 (1.68)
  GAD Follow-up | 0.9 (1.17) | 1.2 (1.55)

8. Secondary Outcome: Depression Assessed by the Patient Health Questionnaire PHQ-2
Description: Patient Health Questionnaire is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of not at all, several days more than half the days, and-nearly every day, respectively. Total score for the two ranges from 0 to 6 with higher number worse depression outcome.
Time Frame: Baseline to 2 week follow up
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on PHQ-2 scale
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Number analyzed (Participants) | 23 | 11
score on PHQ-2 scale
  Change in PHQ (Follow up-Baseline) | -1.10 (1.34) | 0 (0.47)
  PHQ Baseline | 2 (1.53) | 1.33 (1.44)
  PHQ Follow-up | 0.86 (1.39) | 1.3 (1.7)

9. Secondary Outcome: Short Form Health Survey (SF12v12)
Description: Health-related quality of life assessment Short Form Health Survey 12 has two composite scores (Physical composite score and Mental composite score). Each score has a range of 0 to 100 with higher scores indicating better health outcomes.
Time Frame: Baseline to 2 week follow up
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on SF 12 scale
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Number analyzed (Participants) | 23 | 11
score on SF 12 scale
  Change in Physical Score (Follow-up- Baseline) | 7.3 (6.42) | -1.85 (6.81)
  Physical Score Baseline | 27.0 (6.87) | 29.1 (4.80)
  Physical Score Follow up | 27.9 (8.61) | 27.7 (7.22)
  Change in Mental Score (Follow-up - Baseline) | 6.56 (7.25) | 5.65 (7.89)
  Mental Score Baseline | 43.6 (12.3) | 43.5 (13.1)
  Mental Score Follow up | 50.4 (10.2) | 48.6 (16.2)

10. Secondary Outcome: Back Pain Disability Assessed by the Back Pain Oswestry Disability Index (ODI)
Description: Pain Management assessments for patients with back pain. Oswestry Disability Index For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5 with 50 as a highest score; higher scores indicating a worse disability outcome from back pain. Scale is 0-50.
Time Frame: Baseline to 2 week follow up
Population: For the VR-GI group, 9 participants out of the 12 participants with a CBP diagnosis were analyzed as 1 participant did not receive intervention, 1 participant discontinued intervention, and 1 did not complete a post-intervention questionnaire. For the AO-GI group, 6 participants were analyzed as they had a CBP diagnosis.
Measure: Mean (Standard Deviation); unit: score on Oswestry Disability scale
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Number analyzed (Participants) | 9 | 6
score on Oswestry Disability scale
  Change in ODI (Follow-up - Baseline) | -3.44 (3.40) | -4.83 (7.65)
  ODI Baseline | 24.6 (5.66) | 25.8 (8.98)
  ODI Follow up | 20.8 (5.65) | 21 (9.07)

11. Secondary Outcome: Complex Regional Pain Syndrome Symptoms Assessed by the CSS 17 Patientobservation Portion
Description: Pain management assessments for patients with CRPS. Complex Regional Pain Syndrome (CRPS) Severity Score (CSS-17) 0 absence of symptoms, 1 presence of symptoms, 0-8, higher score indicate worse symptom outcome.
Time Frame: Baseline to 2 week follow up
Population: CSS-17 was unreported due to participants receiving an incomplete CSS-17 questionnaire.
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Daily Pain Numerical Rating Scale
Description: Rating of current pain intensity from 0-10 with higher number indicated worse pain outcomes
Time Frame: Baseline to 2 week follow up
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: difference score on pain scale
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
Number analyzed (Participants) | 23 | 12
difference score on pain scale
  Change in Pain Score (Follow-up - Baseline) | -0.906 (0.851) | -.757 (0.489)
  Pre Pain Score | 5.75 (1.5) | 5.49 (1.41)
  Post pain Score | 4.82 (1.48) | 4.8 (1.47)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: For the VR-GI group, adverse events were calculated with 23 participants as one participant did not receive allocated intervention.
Arm/Group | Virtual Reality Guided Imagery (VR-GI) | Audio Only Guided Imagery (AO-GI)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/12
Other Adverse Events (participants affected / at risk) | 5/23 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Virtual Reality Guided Imagery (VR-GI) (N=23) | Audio Only Guided Imagery (AO-GI) (N=12)
device usage (Product Issues) | 5 (5) | 0 (0) — difficulty using device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT04849897/Prot_SAP_001.pdf